CLINICAL TRIAL: NCT06756906
Title: Comparison of the Effects of High Flow Nasal Oxygen and Standard Nasal Oxygen Therapy in Preventing Hypoxia in Minor and Moderate Burn Patients Treated Under Sedation
Brief Title: Comparison of High Flow Nasal Oxygen and Nasal Cannula in Burn Patients Under Sedation
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Cihan Döğer, Assoc. Prof. MD, Ankara City Hospital Bilkent
Other Study IDs: E2-24-6462
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Burn Injury; Hypoxia; Sedation
Keywords: HFNO; Sedation; burn injury
MeSH Terms: conditions — Burns; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Standard nasal oxygen therapy: Patients will be preoxygenated with 8L/min oxygen and will receive 3L/min oxygen throughout the procedure.
- Group 2: High-flow nasal oxygen therapy (HFNO): Patients who will receive HFNO will be preoxygenated with HFNO 40 l/min with FiO2 100% 3 min before induction. Patients will receive HFNO 50 l/min with FiO2 50% throughout the procedure.

SUMMARY:
Burn-related pain is severe and often difficult to manage. Burn patients often require high doses of opioids and anxiolytics. Anesthetic agents used during sedation such as benzodiazepines, propofol and opioids can cause respiratory depression, predisposing patients to hypoventilation and hypoxemia due to airway obstruction. Oxygen is administered to patients with a standard nasal cannula during sedation. High Flow Nasal Oxygen (HFNO) helps to improve the oxygenation of patients with respiratory distress by delivering high flow humidified oxygen through the nasal cannula at a high rate of up to 40-70 liters per minute. The aim of this study was to compare the effects of HFNO and nasal oxygen therapy in preventing hypoxemia in deeply sedated burn patients.

DETAILED DESCRIPTION:
This research is an observational prospective case-control study conducted in the Burns Center of Ankara Bilkent City Hospital. The aim of the study was to compare standard nasal oxygen therapy with High Flow Nasal Oxygen (HFNO) therapy in terms of hypoxemia in patients undergoing surgery for minor and moderate burns under deep sedation. Volunteer patients over 18 years of age, in the ASA (American Society of Anesthesiology) I-III risk group, who will undergo burn operation will be included in the study. Patients will be informed about the scope of the study, possible risks and benefits before participating in the study, and informed consent will be obtained from all participants by signing the informed consent form.

A total of 70 patients will be included in the study. The study consists of 2 groups. Group 1: Standard nasal oxygen (n:35), Group 2: HFNO (n:35) Before starting induction, patients who will be given nasal oxygen will be preoxygenated with 100% oxygen for 3 min with an oxygen flow rate of 8 l/min. Patients who will receive HFNO will be preoxygenated with HFNO 40 l/min with FiO2 100% 3 min before induction. Patients will be premedicated with 1 mg iv midazolam and 1 mcg/kg fentanyl 1 min before induction. During the induction phase, 1% propofol-ketamine (0.5-1 mg/kg) will be administered and an additional dose of propofol-ketamine will be administered according to the patient's BIS value and the total drug dose will be noted. Non-invasive arterial blood pressure, heart rate, electrocardiogram (ECG), oxygen saturation, SpO2, BIS and NIRS values will be recorded before and every 5 minutes during the procedure. Patient demographics, total procedure time, amount of anesthetic agent used, heart rate and other clinical parameters will also be recorded. Ramsey sedation scale of the patients during the procedure and Aldrete scores at the end of the procedure will be evaluated. In case of apnea or desaturation, maneuvers such as patient stimulation, chin lifting, or increasing oxygen flow were performed and recorded.

The statistical package program SPSS 25.0 (Armonk, NY: IBM Corp.) will be used for data analysis. Descriptive statistics (frequency, percentage, minimum, maximum, mean, standard deviation, median, min-max, IQR) will be used. Pearson chi-square test, Fisher or Yates x2 tests will be used to compare qualitative data. The conformity of the data to normal distribution will be evaluated by Kolmogorov-Smirnov and Shapiro-Wilk tests, skewness-kurtosis and graphical methods (histogram, Q-Q Plot, Stem and Leaf, Boxplot). For normally distributed quantitative data, independent samples t test or one way ANOVA will be applied. For non-normally distributed data, Mann-Whitney U test or Kruskal-Wallis test will be used. Paired t test or Friedman test will be used to compare repeated measures. The relationship between variables will be evaluated by Pearson or Spearmans's Rho Correlation test. P<0.05 will be accepted as statistical significance level.

ELIGIBILITY:
Inclusion Criteria : Voluntary patients over 18 years of age -ASA(American Society of Anaesthesiologists) I-III risk scores Exlusion Criteria

Exclusion Criteria:

* Intubation
* Tracheostomies
* Need for oxygen therapy due to preexisting disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for burn treatment under sedation in Ankara City Hospital's Burn Center will be included
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-01-27 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation SpO2 levels of the cases in % | Oxygen saturation levels will be recorded before induction and every 5 minutes throughout the procedure.
  Each patient will be monitored with an oxygen saturation probe and SpO2 levels of the cases will be recorded before induction of sedation and every 5 minutes, throughout the procedure. Hypoxemia will be detected.

SECONDARY OUTCOMES:
Number of interventions over procedure time | Number of maneuvers performed throughout the procedure.
  In case of apnea or desaturation, airway interventions will be performed and recorded throughout the procedure.

OTHER OUTCOMES:
Systolic, diastolic and mean blood pressures will be recorded in mmHg | Blood pressure monitorization will be performed induction and every 5 minutes throughout the procedure.
  Before induction patients will be monitored, and systolic, diastolic and mean blood pressures will be recorded before induction and every 5 minutes throughout the procedure.
Heart beat will be recorded in beats per minute | Heart beat monitorization will be performed before induction and every 5 minutes throughout the procedure.
  Heart beats will be recorded before induction and every 5 minutes throughout the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Erkılıç, Assoc Prof, Principal Investigator — Ankara Bilkent City Hospital, Department of Anesthesiology; Huriye Bilge Tuncer, MD, Principal Investigator — Ankara Bilkent City Hospital, Department of Anesthesiology; Merve Akın, Assoc Prof, Principal Investigator — Ankara Bilkent City Hospital, Department of General Surgery
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Date will be shared after publication of the study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginnning right after publication and ending 2 years after the publication of results
Access Criteria: Data required for research will be shared

REFERENCES:
- [Background] Service JA, Bain JS, Gardner CP, McNarry AF. Prospective Experience of High-flow Nasal Oxygen During Bronchoscopy in 182 Patients: A Feasibility Study. J Bronchology Interv Pulmonol. 2019 Jan;26(1):66-70. doi: 10.1097/LBR.0000000000000533. PMID 30048415
- [Background] Khanna P, Haritha D, Das A, Sarkar S, Roy A. Utility of high-flow nasal oxygen in comparison to conventional oxygen therapy during upper gastrointestinal endoscopic procedures under sedation: A systematic review and meta-analyses. Indian J Gastroenterol. 2023 Feb;42(1):53-63. doi: 10.1007/s12664-022-01308-6. Epub 2023 Feb 13. PMID 36780095
- [Background] Spence EA, Rajaleelan W, Wong J, Chung F, Wong DT. The Effectiveness of High-Flow Nasal Oxygen During the Intraoperative Period: A Systematic Review and Meta-analysis. Anesth Analg. 2020 Oct;131(4):1102-1110. doi: 10.1213/ANE.0000000000005073. PMID 32925331